CLINICAL TRIAL: NCT02782767
Title: Comparison of Continuous Wound Catheter Infusion Versus Continuous Epidural Infusion in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Arun Raja T, Junior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MDTG105
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Upper Gastrointestinal Surgery; Post-operative Analgesia; Wound Infusion Catheter; Upper Midline Incision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural catheter infusion (Active Comparator): epidural catheter in the thoracic vertebra level to provide local anesthetic infusion
  Interventions: Other: Epidural infusion
- Wound catheter infusion (Experimental): A multiorificed wound infusion catheter kept within the incision site to provide continuous local anesthetic infusion
  Interventions: Other: Wound catheter infusion

INTERVENTIONS:
Other: Wound catheter infusion — Wound catheter has multiple holes spread around 360 degrees throughout its active length. It is placed in the musculofascial plane during closure of the wound. Local anaesthetic infusion will be delivered through the catheter.
  Arms: Wound catheter infusion
Other: Epidural infusion — Epidural catheter will be placed in the level T7-T9 , and local anaesthetic infusion will be given
  Arms: Epidural catheter infusion

SUMMARY:
Comparison of efficacy in management of pain in abdominal surgery between epidural versus wound infusion catheter {catheter placed within the incision site}

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I-III , undergoing upper gastrointestinal surgery involving upper midline incision

Exclusion Criteria:

* Refusal to give consent.
* Contraindication to epidural analgesia (e.g.localized sepsis , Raised ICP , Myelopathy , Peripheral neuropathy ,Inherited coagulopathy)
* Addiction to opioids, or alcohol, or history of any other substance abuse.
* Allergy to local anaesthetic drugs.
* Pregnancy.
* Inability to communicate (e.g. known psychiatric disorders)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
NRS (Numerical Rating Score) in the two groups postoperatively | 24 hrs post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arun Raja Thangavel, MBBS, Principal Investigator — Junior Resident , MD Anaesthesia and Intensive care
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided